CLINICAL TRIAL: NCT02046928
Title: A Phase 2 Trial to Determine the Safety, Tolerability, and Efficacy of A6, a CD44 Binding Peptide, for the Treatment of Patients With Chronic Lymphocytic Leukemia
Brief Title: Safety, Tolerability and Efficacy of A6 in Patients With Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Ångstrom Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6-005
Record Dates: First submitted 2014-01-20; First posted 2014-01-28 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; CLL; SLL
Keywords: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A6 (Experimental): A6 is administered subcutaneously two times a day for 6 cycles (1 cycle = 28 days).
  Interventions: Drug: A6

INTERVENTIONS:
Drug: A6 — A6 is self-administered subcutaneously two times a day for 6 cycles (1 cycle = 28 days).

SUMMARY:
This study will assess the efficacy, safety and pharmacodynamic markers of the study drug, A6, in patients with CLL and small lymphocytic lymphoma (SLL).

DETAILED DESCRIPTION:
In patients diagnosed with CLL or SLL, study medication will be injected subcutaneously two times a day in an outpatient setting for up to 6 cycles (28 days = 1 cycle) prior to the primary endpoint assessment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL or SLL based on IWCLL Criteria
* Measurable or evaluable disease based on IWCLL criteria
* Previously untreated patients who have been counseled on approved alternative therapeutic options. Not a candidate for fludarabine/cyclophosphamide/rituximab (FCR) or has preference to not receive chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) status of 0-2.
* Adequate bone marrow, renal, liver, cardiac and pulmonary function.
* Life expectancy of greater than or equal to 6 months.

Exclusion Criteria:

* Receipt of other cancer therapy, immunomodulatory drug therapy or immunosuppressive therapy within 4 weeks prior to 1st dose.
* Receipt of corticosteroids > 20 mg/day within 4 weeks prior to1st dose
* Major surgery or radiation within 4 weeks prior to 1st dose
* Presence of uncontrolled infection requiring systemic therapy
* Active second malignancy other than non-melanoma skin cancer
* Uncontrolled autoimmune anemia or thrombocytopenia
* Receipt of any investigational agent within 4 weeks prior to 1st dose
* Pregnant or lactating female
* Any severe, acute or chronic medical or psychiatric condition, or lab abnormality that may increase the risk associated with trial participation, study drug administration or interfere with informed consent process or compliance with requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Assessed at Day 28 of Cycle 6
  International Workshop on Chronic Lymphocytic Lymphoma (IWCLL) Guidelines for response of clinical, hematological, and bone marrow features.

SECONDARY OUTCOMES:
Safety of A6 | Throughout 6 Cycles (6 months)
  Nature and frequency of adverse events
Determine IWCLL response rate in the Intent-To-Treat Population | Throughout 6 Cycles (6 months)
Determine the response in patients who received all 6 cycles of A6 | 6 months
Determine progression-free survival | Throughout 6 Cycles (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Choi, MD, Principal Investigator — Moores Cancer Center, UCSD
Locations (1):
- Moores Cancer Center, UCSD, La Jolla, California, United States